CLINICAL TRIAL: NCT03716960
Title: The Effects of Pumpkin Seed Oil Supplementation on Vascular Hemodynamics, Stiffness and Cardiac Autonomic Function in Postmenopausal Women.
Brief Title: The Effects of Pumpkin Seed Oil Supplementation on Cardiovascular Function in Postmenopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marymount University (Other)
Responsible Party: Principal Investigator, Alexei Wong, Assistant Professor, Marymount University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 321
Record Dates: First submitted 2018-10-20; First posted 2018-10-23 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Elevated Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pumpkin Seed Oil (Experimental): This arm involved 6 weeks of PSO consumption. Subject were supplemented with 3 g/day of PSO which was ingested in the form of 1g capsules with each main meal of the day (breakfast, lunch and dinner). Likewise,
  Interventions: Other: Pumpkin Seed Oil
- Placebo (Placebo Comparator): This arm involved 6 weeks of placebo consumption. Subject consumed 1 capsule of maltodextrin with each main meal of the day to match the dose and number of capsules ingested daily by the PSO group.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Pumpkin Seed Oil — This intervention consisted of 6 weeks of PSO consumption. Subject were supplemented with 3 g/day of PSO which was ingested in the form of 1g capsules with each main meal of the day (breakfast, lunch and dinner).
  Arms: Pumpkin Seed Oil
Other: Placebo — This intervention consisted of 6 weeks of placebo consumption. Subject consumed 1 capsule of maltodextrin with each main meal of the day to match the dose and number of capsules ingested daily by the PSO group.
  Arms: Placebo

SUMMARY:
Postmenopausal women have a higher prevalence of cardiovascular (CV) disease than age-match men. Growing evidence from rat studies have demonstrated CV-protective effects of pumpkin seed oil (PSO).

The investigators hypothesis is that PSO would improve CV health in postmenopausal women.

DETAILED DESCRIPTION:
The purpose of the study is to examine the effects of 6 weeks of PSO on arterial and autonomic function in postmenopausal women. Specific aims of the study are to:

To investigate the extent to which PSO will improve cardiovascular disease risk factors by assessing arterial stiffness, aortic BP and wave reflection, and autonomic function (heart rate variability).

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45 to 65 years of age
* At least 1 year after menopause
* BMI <39.9
* Sedentary or low active (less than 2 hr per wk)

Exclusion Criteria:

* known heart disease
* peripheral vascular disease
* diabetes, body mass index
* BMI> 40 kg/m2
* other chronic diseases
* taking medications (e.g., hormone replacement therapy, beta blockers, calcium channel blockers, antidepressants and stimulants) that could affect the outcome variables
* smokers
* history of steady exercise or received exercise training and dietary changes in the last year

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 6 weeks
  Non-invasive measures of brachial and aortic blood pressure
Pressure Wave Reflection | 6 weeks
  Using the augmentation index
Arterial Stiffness | 6 weeks
  Using the stiffness index
Heart rate variability | 6 weeks
  R-R intervals were collected during 6 min using a validated wireless monitor (Polar 800CX; Polar Electro OY, Kempele, Finland) via a chest strap interfaced with a PC. All R-R intervals were inspected for artifacts and premature beats.

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Wong, Ph.D, Principal Investigator — Marymount University
Locations (1):
- Marymount University, Arlington, Virginia, United States

REFERENCES:
- [Derived] Wong A, Viola D, Bergen D, Caulfield E, Mehrabani J, Figueroa A. The effects of pumpkin seed oil supplementation on arterial hemodynamics, stiffness and cardiac autonomic function in postmenopausal women. Complement Ther Clin Pract. 2019 Nov;37:23-26. doi: 10.1016/j.ctcp.2019.08.003. Epub 2019 Aug 8. PMID 31445363